CLINICAL TRIAL: NCT03560622
Title: Functional Neuroimaging Feedback for Focused Ultrasound Thalamotomy for Tremor Surgery
Brief Title: Functional Neuroimaging Feedback for Focused Ultrasound Thalamotomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vibhor Krishna (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Focused Ultrasound Foundation (Other)
Responsible Party: Sponsor-Investigator, Vibhor Krishna, Assistant Professor- Neurological Surgery, Ohio State University
Organization: Ohio State University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018H0035
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Essential Tremor
Keywords: focused ultrasound; fMRI
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Intervention Model Description: Ten adults with refractory ET (ET cohort) and 20 healthy controls (control cohort) will undergo multi-modality neuroimaging (structural imaging, diffusion tensor imaging (DTI), task-based functional MRI (t-fMRI), and resting state functional MRI (rs-fMRI)). In addition the ET cohort will also undergo imaging with the identical protocol immediately after and 24 hours after FUS-T.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ET cohort (Active Comparator): Ten adults with refractory ET (ET cohort) will undergo multi-modality neuroimaging (structural imaging, diffusion tensor imaging (DTI), task-based functional MRI (t-fMRI), and resting state functional MRI (rs-fMRI)). In addition the ET cohort will also undergo imaging with the identical protocol immediately after and 24 hours after FUS-T.
  Interventions: Device: multi-modality neuroimaging
- control cohort (Experimental): Twenty adult healthy controls (control cohort) will undergo multi-modality neuroimaging (structural imaging, diffusion tensor imaging (DTI), task-based functional MRI (t-fMRI), and resting state functional MRI (rs-fMRI)).
  Interventions: Device: multi-modality neuroimaging

INTERVENTIONS:
Device: multi-modality neuroimaging — multi-modality neuroimaging consists of structural imaging, diffusion tensor imaging (DTI), task-based functional MRI (t-fMRI), and resting state functional MRI (rs-fMRI).

SUMMARY:
Focused ultrasound for Essential Tremor is an FDA approved treatment performed by neurosurgeons at the Ohio State Center for Neuromodulation that utilizes ultrasound technology to create a lesion in the thalamus of Essential Tremor patients. In order to improve long term effectiveness and reduce potential for side effects, brain imaging may be used to examine the functional connectivity of certain brain networks during the procedure. In order to investigate functional connectivity changes with these long term goals in mind, in this study neuroimaging will be taken immediately before, immediately after, and 24 hours after the focused ultrasound procedure for 10 Essential Tremor patients. One series of neuroimaging will also be conducted for 20 healthy control subjects to serve as a comparison. This study will not introduce any risks above standard of care, and may lead to improved long term outcomes of patients undergoing the Focused Ultrasound procedure.

DETAILED DESCRIPTION:
To calculate the connectivity correlates of tremor (CCT) by analyzing and comparing functional connectivity in the tremor network in ET patients and healthy controls. The fMRI data will be acquired in two separate conditions: t-fMRI and rs-fMRI. a. For t-fMRI, patients will perform simple repetitive tasks (e.g. finger tapping, hand grasping) to identify activation clusters within tremor network. Functional connectivity between the clusters will be calculated by creating cross-correlation matrices. A sensitivity analysis will then be performed to determine an optimal value of CCT to distinguish ET patients from controls. b. For rs-fMRI the hubs within tremor network will be identified with a state-of-the-art multimodality atlas. Cross-correlation matrices will be created to calculate measures of functional connectivity. A sensitivity analysis will then be performed to determine an optimal value of CCT to distinguish ET patients from controls. 2. To study changes in functional connectivity in the tremor network before, immediate postoperative and and 24-hours after FUS-T in ET patients. a. The CCT will be calculated and compared between baseline, immediate postoperative and 24-hours post-operative conditions to determine the effect of FUS-T. For this sub-aim the connectivity data will be separately analyzed for t-fMRI and for rs-fMRI. b. The CCT in immediate postoperative and 24-hours post-operative condition among ET patients will be compared to healthy controls to determine whether FUS-T restored the abnormal connectivity in tremor network. For this sub-aim the connectivity data will be separately analyzed for t-fMRI and rs-fMRI.

ELIGIBILITY:
Inclusion Criteria:

* The tremor diagnosis, disability and medically refractory status are agreed upon by at least two movement disorder trained physicians (neurologists and/or neurosurgeons).
* The patient is deemed suitable for surgical therapy for tremor with VIM targeting.
* The patient is willing to participate in the study and provides written informed consent.
* The patient is able to clearly communicate clinical findings with the clinical team.
* The patient is willing to participate in at least one follow-up visit at 3 or 6 months.
* In order to maintain uniformity of image acquisition only patients undergoing imaging with the 3T MRI at The Ohio State University Wexner Medical Center will be included.

Exclusion Criteria:

* Medically unstable - uncontrolled hypertension, coronary artery disease, significant pulmonary problems, active history of bleeding disorders or anticoagulation.
* Other diagnoses of tremor like Parkinson's disease, traumatic tremor, dystonic tremor, and/or tremor associated with multiple sclerosis
* Unwilling or unable to undergo awake tremor surgery.
* Tremor patients undergoing surgery with targets other than the VIM.
* Significant motion artifact in imaging.
* Unable to undergo 3T MRI imaging.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
connectivity correlates of tremor (CCT) | during the surgical procedure
  CCT will be calculated by analyzing and comparing functional connectivity in the tremor network in ET patients and healthy controls. The fMRI data will be acquired in two separate conditions: t-fMRI and rs-fMRI. Both t-fMRI and rs-MRI will be calculated based upon functional connectivity between the dentate nucleus, ventral intermediate nucleus, globus pallidus, motor and premotor cortex sensitivity analysis will then be performed to determine an optimal value of CCT to distinguish ET patients from controls.

SECONDARY OUTCOMES:
changes in functional connectivity | immediately post-operative and 24-hours after surgery for ET patients
  2. To study changes in functional connectivity in the tremor network before, immediate postoperative and and 24-hours after FUS-T in ET patients.
  1. The CCT will be calculated and compared between baseline, immediate postoperative and 24-hours post-operative conditions to determine the effect of FUS-T. For this sub-aim the connectivity data will be separately analyzed for t-fMRI and for rs-fMRI.
  2. The CCT in immediate postoperative and 24-hours post-operative condition among ET patients will be compared to healthy controls to determine whether FUS-T restored the abnormal connectivity in tremor network. For this sub-aim the connectivity data will be separately analyzed for t-fMRI and rs-fMRI.

CONTACTS AND LOCATIONS:
Overall Officials: Vibhor Krishna, MD SM, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State Medical Center, Columbus, Ohio, United States